CLINICAL TRIAL: NCT06288542
Title: The Relationship of Preoperative Intravenous Dextrose Infusion to Postoperative Nausea and Vomiting in Gynecological Laparoscopic and Hysteroscopic Surgeries: A Randomized Control Trial
Brief Title: Preoperative Dextrose Infusion and Postoperative Nausea and Vomiting
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmin Hassab elnaby, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MD-250-2022
Record Dates: First submitted 2024-02-25; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Effect of Dextrose on Postoperative Nausea and Vomiting
Keywords: dextrose infusion; postoperative nausea and vomiting; gynecological laparoscope and hysteroscope
MeSH Terms: conditions — Vomiting; Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group c (No Intervention): control group . this group will not receive any iv fluids
- group d (Experimental): Group D will receive 1 mL/kg/h 5% Dextrose infusion, applied preoperatively during fasting until induction of anesthesia
  Interventions: Other: group d
- group r (Active Comparator): this group will receive 1 mL/kg/h ringer infusion, applied preoperatively during fasting until induction of anesthesia
  Interventions: Other: group R

INTERVENTIONS:
Other: group d — this group will receive 1 mL/kg/h 5% Dextrose infusion, applied preoperatively during fasting until induction of anesthesia
  Other Names: dextrose group
  Arms: group d
Other: group R — this group will receive 1 mL/kg/h ringer infusion, applied preoperatively during fasting until induction of anesthesia
  Other Names: ringer group
  Arms: group r

SUMMARY:
This research aims to investigate the efficacy of preoperative intravenous infusion of dextrose 5% during fasting in lowering the incidence and severity of post-operative nausea and vomiting related to laparoscopic gynaecologic procedures

DETAILED DESCRIPTION:
A history of PONV risk factors will be recorded. After consenting, patients will be assigned using a computerized randomization function to Ringer solution (group R) or 5% dextrose (group D) or control group (group C). Group D will receive 1 mL/kg/h 5% Dextrose infusion, applied preoperatively during fasting until induction of anesthesia. Group R will receive 1 mL/kg/h ringer infusion, applied preoperatively during fasting until induction of anesthesia. Group C will receive no fluids. The anesthesia providers, surgeons, perioperative nurses, postanesthesia care unit (PACU) nurses and investigators will be blinded to group assignment throughout.

As for pre-medication, all patients will receive IV midazolam (0.02 mg/kg). Anesthesia will be induced with propofol (1.5-2 mg/kg), fentanyl (1-2 μg/kg) and atracurium(o.5mg/kg) to facilitate endotracheal intubation. The lungs will be mechanically ventilated and anesthesia will be maintained with isoflurane in O2/air. Intraoperative IV maintenance fluid will be standardized at 3 mL/kg/h with additional IV crystalloid given as needed at the discretion of the anesthesia provider if arterial blood pressure decreased >20% from baseline. For postoperative pain relief, paracetamol 1 g will be given I.V. during surgery in all patients and continued orally after operation (1g every 6 h). In addition, all patients will be ambulated within 6 h after completion of surgery. Standardized antiemetic and analgesic rescue medications will be available. Patients will receive no rescue antiemetic medication when the VRS score is 0 to 2; 1 dose of rescue medication when the VRS score is 3 to 6; and ≥2 doses for nausea score of 7 to 10, to reduce the nausea score to 0 to 2.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients scheduled for elective laparoscopic gynecological/hysteroscopic procedures will be considered for inclusion
* ASA physical status I and ll.

Exclusion Criteria:

* patients with a previous history of PONV.
* Patients with motion sickness, coagulopathy, diabetes mellitus, or severe hypertension
* patients with cardiac, renal or hepatic dysfunction.
* patients receiving an antiemetic agent within 24 h before surgery or cases where complications occurs during the surgery
* patients who have abnormal blood glucose on the night before surgery
* patients who are unable to understand and use the verbal rating scale (VRS);Growth developmental, and motor-mental retardation.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
frequency of post-opertive nausea and vomiting in 24 hour | FROM ENROLLMENT TO 24 HOURS AFTER SURGERY
  using verbal rating scale (VRS)

SECONDARY OUTCOMES:
TOTAL AMOUNT OF ANTIEMETIC REQUIRED | From end of surgery to 24 hours postoperative